CLINICAL TRIAL: NCT00240448
Title: A Randomised, Double-blind, Double-dummy, Placebo-controlled, Forced-titration, Comparison of MICARDIS® HCT (Telmisartan 80 mg / Hydrochlorothiazide 25 mg) Versus DIOVAN® HCT (Valsartan 160 mg / Hydrochlorothiazide 25 mg) Using Seated Trough Cuff Blood Pressure in Patients With Stage 1 and Stage 2 Hypertension
Brief Title: A Randomized, Double-blind, Placebo Controlled Comparison of Telmisartan Hydrochlorothiazide (HCT) and Valsartan HCT in Hypertension (HTN) Stage I/II Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.421
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Hydrochlorothiazide; Valsartan

INTERVENTIONS:
Drug: telmisartan 80 mg/hydrochlorothiazide 25 mg
Drug: valsartan 160 mg/hydrochlorothiazide 25 mg
Drug: placebo

SUMMARY:
The primary objective of this study is to compare the effectiveness of telmisartan 80 mg/hydrochlorothiazide 25 mg [Micardis HCT] to valsartan 160 mg/hydrochlorothiazide 25 mg [Diovan HCT] and placebo in the treatment of Stage 1 and Stage 2 hypertension.

ELIGIBILITY:
Inclusion criteria

1. Ability to provide written informed consent.
2. Age 18 years or older.
3. Ability to stop current antihypertensive therapy without unacceptable risk to the patient (investigator's discretion).
4. Seated cuff DBP of 95 mmHg at Visit 2 (baseline).

Exclusion criteria

1. Pre-menopausal women (last menstruation 1 year prior to start of run-in period) who:

   * Are not surgically sterile and/or
   * Are nursing or pregnant
   * Are of child-bearing potential and are NOT practicing acceptable means of birth control, do NOT plan to continue using this method throughout the study and do NOT agree to submit to periodic pregnancy testing during participation in studies of > 3-months duration. Acceptable methods of birth control include oral, implantable, transdermal, or injectable contraceptives, and Intra-Uterine Device (IUD).
2. Known or suspected secondary hypertension.
3. Mean seated SBP >= 180 mmHg or mean seated DBP >= 120 mmHg during any clinic visit prior to randomization.
4. Hepatic and/or renal dysfunction as defined by the following laboratory parameters:

   * SGPT (ALT) or SGOT (AST) > 2 times the upper limit of normal range, or
   * Serum creatinine > 3.0 mg/dL or creatinine clearance < 0.6 ml/sec.
5. Bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, post-renal transplant or with only one kidney.
6. Clinically relevant hypokalemia or hyperkalemia.
7. Uncorrected volume depletion.
8. Uncorrected sodium depletion.
9. Primary aldosteronism.
10. Hereditary fructose intolerance.
11. Biliary obstructive disorders, cholestasis or moderate to severe hepatic insufficiency.
12. Patients who have previously experienced symptoms characteristic of angioedema during treatment with ACE inhibitors or angiotensin II receptor antagonists.
13. History of drug or alcohol dependency within six months prior to start of run-in period.
14. Chronic administration of any medications known to affect blood pressure, etc.
15. Any investigational drug therapy within one month of start of run-in period.
16. known hypersensitivity to any component of the formulation study drugs (telmisartan, valsartan, HCT).
17. Contra-indication to a placebo run-in period (e.g. stroke within the past six months, MI, cardia surgery, PTCA or angina within the past three months prior to the start of run-in period.
18. Any other clinical condition which, in the opinion of the principal investigator, would not allow safe completion of the protocol and safe administration of telmisartan, valsartan, or HCT.
19. Night shift workers.
20. Clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the investigator.
21. NYHA functional class CHF III-IV.
22. Hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of aortic or mitral valve.
23. Patients whose diabetes has been unstable and uncontrolled for at least the past 3 months as defined by a HbA1c >/= 10%.
24. Concomitant use of lithium or cholestyramine or colestipol resins (potential drug interactions with HCT).
25. History of non-compliance with prescribed medication or protocol procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1109 (Actual)
Dates: Start 2003-09; Primary Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean seated trough cuff diastolic and systolic blood pressure measurements at the end of an 8-week treatment period

SECONDARY OUTCOMES:
Percentage of responders based on change from baseline in cuff diastolic and systolic blood pressure measurements at the end of an 8-week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (100):
- United States (100):
  - Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - Boehringer Ingelheim Investigational Site, Sctoosdale, Arizona
  - Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - Boehringer Ingelheim Investigational Site, Bentonville, Arkansas
  - Boehringer Ingelheim Investigational Site, Carlisle, Arkansas
  - Boehringer Ingelheim Investigational Site, Hot Springs, Arkansas
  - Boehringer Ingelheim Investigational Site, Concord, California
  - Memorial Research Medical Clinic, Long Beach, California
  - Boehringer Ingelheim Investigational Site, Orange, California
  - Boehringer Ingelheim Investigational Site, Riverside, California
  - Clinical Trials Research, Roseville, California
  - Boehringer Ingelheim Investigational Site, Sacramento, California
  - Boehringer Ingelheim Investigational Site, San Leandro, California
  - Boehringer Ingelheim Investigational Site, Santa Ana, California
  - Boehringer Ingelheim Investigational Site, Sepulveda, California
  - Boehringer Ingelheim Investigational Site, Spring Valley, California
  - Boehringer Ingelheim Investigational Site, Torrance, California
  - Boehringer Ingelheim Investigational Site, Boulder, Colorado
  - Boehringer Ingelheim Investigational Site, Bridgeport, Connecticut
  - Boehringer Ingelheim Investigational Site, Farmington, Connecticut
  - Clinical Research Consultants, Inc., Trumbull, Connecticut
  - Boehringer Ingelheim Investigational Site, Waterbury, Connecticut
  - Boehringer Ingelheim Investigational Site, Newark, Delaware
  - Boehringer Ingelheim Investigational Site, Coral Gables, Florida
  - Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - Boehringer Ingelheim Investigational Site, Fort Myers, Florida
  - Boehringer Ingelheim Investigational Site, Holiday, Florida
  - Boehringer Ingelheim Investigational Site, Hollywood, Florida
  - Christopher Chappel, MD, Kissimmee, Florida
  - Boehringer Ingelheim Investigational Site, Largo, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Boehringer Ingelheim Investigational Site, Palm Harbor, Florida
  - Boehringer Ingelheim Investigational Site, Panama City, Florida
  - Attention: Larry I. Gilderman, D.O., Pembroke Pines, Florida
  - Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - Grady Memorial Hospital, Atlanta, Georgia
  - Boehringer Ingelheim Investigational Site, Conyers, Georgia
  - Treasure Valley Cardiology, Boise, Idaho
  - Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Herron Medical Center, Ltd., Chicago, Illinois
  - Boehringer Ingelheim Investigational Site, Orland Park, Illinois
  - N Touch Research, Peoria, Illinois
  - Midwest Institute for Clinical Research Inc., Indianapolis, Indiana
  - Boehringer Ingelheim Investigational Site, Waterloo, Iowa
  - Boehringer Ingelheim Investigational Site, Shawnee, Kansas
  - Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - Attn:William Smith, New Orleans, Louisiana
  - Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - Boehringer Ingelheim Investigational Site, Brookline, Massachusetts
  - Waltham Hospital, Waltham, Massachusetts
  - Boehringer Ingelheim Investigational Site, Troy, Michigan
  - Boehringer Ingelheim Investigational Site, Brooklyn Center, Minnesota
  - Radiant Research, Edina, Minnesota
  - Boehringer Ingelheim Investigational Site, Jackson, Mississippi
  - Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - Department of Medicine, Camden, New Jersey
  - Boehringer Ingelheim Investigational Site, Cherry Hill, New Jersey
  - Boehringer Ingelheim Investigational Site, Kingston, New York
  - Northport VAMC - Medical Service (111), Northport, New York
  - Boehringer Ingelheim Investigational Site, Rochester, New York
  - Boehringer Ingelheim Investigational Site, Scarsdale, New York
  - Boehringer Ingelheim Investigational Site, The Bronx, New York
  - Boehringer Ingelheim Investigational Site, Burlington, North Carolina
  - Boehringer Ingelheim Investigational Site, Cary, North Carolina
  - Boehringer Ingelheim Investigational Site, Durham, North Carolina
  - Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - Boehringer Ingelheim Investigational Site, Stateville, North Carolina
  - Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - Radiant Reseach, Cincinnati, Ohio
  - Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - Ohio State University, Columbus, Ohio
  - Radiant Research, Columbus, Ohio
  - Boehringer Ingelheim Investigational Site, Mansfield, Ohio
  - Boehringer Ingelheim Investigational Site, Mogadore, Ohio
  - Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - Bock Clinical Research, Collegeville, Pennsylvania
  - Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - Boehringer Ingelheim Investigational Site, Pottstown, Pennsylvania
  - Boehringer Ingelheim Investigational Site, East Providence, Rhode Island
  - Boehringer Ingelheim Investigational Site, Greer, South Carolina
  - Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - Boehringer Ingelheim Investigational Site, Austin, Texas
  - Boehringer Ingelheim Investigational Site, Carrollton, Texas
  - Boehringer Ingelheim Investigational Site, Dallas, Texas
  - Boehringer Ingelheim Investigational Site, Houston, Texas
  - Boehringer Ingelheim Investigational Site, McKinney, Texas
  - Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - Clinical Research Center of N. VA, Falls Church, Virginia
  - Boehringer Ingelheim Investigational Site, Lacey, Washington
  - Boehringer Ingelheim Investigational Site, Lakewood, Washington
  - Boehringer Ingelheim Investigational Site, Madison, Wisconsin
  - Boehringer Ingelheim Investigational Site, Milwaukee, Wisconsin